CLINICAL TRIAL: NCT04656548
Title: A Comparative, Retrospective Chart Review of Intended Dwell Time of a PICC Line
Status: Completed | Type: Observational
Sponsor: Access Vascular Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN 20-001
Record Dates: First submitted 2020-12-01; First posted 2020-12-07 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Peripheral ICC; PICC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- HydroPICC: Cohort who received the HydroPICC
  Interventions: Device: HydroPICC
- Standard of Care: Cohort who received something different than HydroPICC

INTERVENTIONS:
Device: HydroPICC — PICC lines
  Other Names: Standard of Care
  Groups: HydroPICC

SUMMARY:
This is a retrospective, matched pair comparative post market review of 4Fr Single Lumen PICC lines. The subjects will be matched by the timeframe of when the HydroPICCs were inserted.

DETAILED DESCRIPTION:
Subjects would have received a 4 Fr Single Lumen PICC line between Aug 2020 and Oct 2020.

The two groups will be HydroPICCs and the standard of care for the facility.

A comparison of multiple endpoints will be evaluated between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been inserted with the HydroPICC during a specific time range.
* During the same time period, any competitor 4 Fr single lumen placed.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients at the study site that received a 4 Fr single lumen PICC line from Aug 2020 through Oct 2020.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Intended dwell time based on a comparison of the actual dwell time to the intended time | August 2020 through October 2020
  Comparison of actual vs intended dwell times of each arm

SECONDARY OUTCOMES:
Comparison of failure rates | August 2020 through October 2020
  Compare the failure rates between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bunch, Principal Investigator — ProVasc
Locations (1):
- Joseph Bunch, Romeoville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No